CLINICAL TRIAL: NCT00802425
Title: Efficacy of AM-111 in Patients With Acute Sensorineural Hearing Loss: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled, Dose-Escalation Phase II Study
Brief Title: Efficacy of AM-111 in Patients With Acute Sensorineural Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auris Medical AG (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-111-CL-08-01; EudraCT number 2008-000132-40
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Hearing Loss
Keywords: Sudden hearing loss; Sudden deafness; Acoustic trauma; Noise trauma
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sudden; Hearing Loss, Noise-Induced | interventions — D-JNKI-1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): AM-111 low dose
  Interventions: Drug: AM-111
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 3 (Experimental): AM-111 high dose
  Interventions: Drug: AM-111

INTERVENTIONS:
Drug: AM-111 — single intratympanic injection
  Arms: 2; 3
Drug: placebo — single intratympanic injection
  Arms: 1

SUMMARY:
The purpose of the study is to determine whether AM-111 is effective in the treatment of acute inner ear hearing loss (acute sensorineural hearing loss, ASNHL).

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral acute sensorineural hearing loss (ASNHL) with onset 48 hours or less ago
* Mean earing loss compared with the unaffected contralateral ear of at least 30 dB in the 3 most affected contiguous frequencies
* Age ≥ 18 years and ≤ 60 years
* Negative pregnancy test for women of childbearing potential
* Able to attend the on-study visits
* Written informed consent before participation in the study

Exclusion Criteria:

* Bilateral ASNHL, if not resulting from acoustic trauma
* Suspected perilymph fistula or membrane rupture
* Barotrauma
* Average air bone gap higher than 20 dB in 3 contiguous frequencies
* History of Meniere disease, autoimmune hearing loss, radiation-induced hearing loss, endolymphatic hydrops, suspected retro-cochlear lesion or fluctuating hearing loss
* Previous ASNHL incident within the past 6 weeks
* Evidence of acute or chronic otitis media or otitis externa on examination
* Any drug-based therapy for inner ear hearing loss that is ongoing or was performed in the past 2 weeks
* Any ongoing or planned concomitant medication for the treatment of tinnitus until 30 days after administration
* Any therapy known as ototoxic (e.g. aminoglycosides, cisplatin, loop diuretics, quinine etc.) in the past 6 months prior to study inclusion
* History of drug abuse or alcoholism
* Any clinically relevant respiratory, cardiovascular, neurological (except vertigo or tinnitus), or psychiatric disorders
* Known hypersensitivity, allergy or intolerance to the study medication or any history of severe abnormal drug reaction
* Women who are breast-feeding, pregnant or who plan a pregnancy during the trial
* Women of childbearing potential who declare being unwilling or unable to practice contraception such as combined oral contraceptives, injectables, hormonal intra-uterine devices, vasectomised partner or sexual abstinence
* Concurrent participation in another clinical trial or participation in another clinical trial within 30 days prior to study entry
* Any current anticoagulant therapy (e.g. Aspirin, Marcumar, etc)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hearing loss | 7 days
  Average change in hearing loss in dB between the baseline and D7 for the three contiguous frequencies with the worst hearing loss, identified at study entry

SECONDARY OUTCOMES:
Hearing loss | Days 3, 30, 90
  Average change in hearing loss in dB between the baseline and D3, D30, and D90 for the three contiguous frequencies with the worst hearing loss, identified at study entry

CONTACTS AND LOCATIONS:
Overall Officials: Markus M Suckfüll, MD, Study Director — LMU Munich
Locations (1):
- LMU Munich Klinikum Grosshadern, Munich, Germany